CLINICAL TRIAL: NCT05221060
Title: Reliability and Validity Study of Urdu Version of Kujala Questionnaire
Brief Title: Urdu Version of Kujala Questionnaire: A Reliability and Validity Study
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-0239
Record Dates: First submitted 2022-02-01; First posted 2022-02-02 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Patellofemoral Pain Syndrome; Anterior Knee Pain Syndrome
Keywords: Kujala Questionnaire; patello femoral pain syndrome; anterior knee pain; validity; functional limitations; reliability
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this research is to interpret and make Kujala Questionnaire adaptable culturally into Urdu to investigate its validity and reliability in Pakistani population among anterior knee pain or patello femoral knee pain. Also check its correlation with 36-Item Short Form Health Survey questionnaire, Lysholm Knee Scoring Scale and 2000 International Knee Documentation Committee Subjective Knee Evaluation Form.

DETAILED DESCRIPTION:
The original English version of Kujala Questionnaire will be translated and culturally adapted as per previous recommendation. In patients with anterior knee pain or patella femoral knee pain, Kujala Questionnaire-Urdu will be distributed among hundred participants choose a convenience sampling technique based on pre-defined inclusion and exclusion criteria. To test reliability of inter/intra observer of ultimate final Urdu Version of Kujala, 36-Item Short Form Health Survey questionnaire, Lysholm Knee Scoring Scale and 2000 International Knee Documentation Committee Subjective Knee Evaluation Form will be filled from patients on the equivalent day, by 2 different bystanders, and for inter observer valuation, with an interval of 30 minutes between the first and second application. Third assessment will be carried out after 7 days of the Observer -1 (re-testing), for intra-observer assessment. Data will be entered and analyzed Cronbach alpha value. Test-retest reliability will be assessed using an intraclass correlation coefficient. Urdu Version of Kujala was evaluated for content validity, construct validity, criterion validity and responsiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders
2. Ages range from 18-40 years
3. They have clinically diagnosed with patello femoral pain syndrome (the diagnosis was established by a positive patellar grind test and pain on touch sensation, found in medial and lateral patellar facets)
4. Participants who acquire 40 to 80 score on Kujala patellofemoral questionnaire before the treatment start
5. Patients willing to participate.

Exclusion Criteria:

1. Participants of the study who has gone through any treatment protocol curative measure for patellofemoral pain syndrome during the last 3 months.
2. Any indication or medical record of lower extremity fracture or surgical procedure
3. History of certain chronic disease e.g. Diabetes Mellitus
4. Participants unable to understand Urdu Version of Kujala

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pakistani population with patello femoral pain syndrome and anterior knee pain.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Kujala Questionnaire | 1st day
  The Kujala Score is mainly used for the patients with anterior knee pain specially patients with patellofemoral pain syndrome that compromises of 13 questions asking about limping, supporting, walking , stairs descent and ascent movement, squat performance, running , jumping , sitting for a long time with flexed knee, pain intensity, swelling around joint, abnormally random knee cap movement that is also called as subluxation of patella ,weakness and atrophy of thigh muscles and lastly about the deficiencies that occurs during flexion movement. Kujala Score ranges from 0 to 100 .The lowest the score, the greater the severity of functional limitations and pain intensity and vice versa.
36-Item Short Form Health Survey Questionnaire | 1st day
  36-Item Short Form Health Survey questionnaire that is self-administered and is largely used for overall health condition and assessment moreover widely used for research purpose. It contains 36 questions, including almost all basic 8 domains like; physical functioning, limitations due to the physical problems, bodily pain, general health perception, social functioning, vitality, limitations due to emotional problems, overall mental health and one more question about any health transition occurred in the last few days. Score ranges from up to 100, higher score means higher level of perfection of general health a low score means the increase level of functional deficit
The Lysholm Score | 1st day
  The Lysholm Score is one of the most common questionnaire used for assessment of severity of pain and level of functional limitations in patients with patellofemoral pain syndrome. The point of concern are the ligaments Injury or mishap to ligament of the knee. Higher scores indicate a better outcome with fewer symptoms or disability.
International Knee Documentation Committee Subjective Knee Evaluation Form | 1st day
  The International Knee Documentation Committee was formulated in 1987 as an International documentation system for knee deficits. Consisting 18 items out which 7 for symptoms, 1 for sports participation, 9 items for Activities of Daily Livings and lastly 1 for the current knee situation and function. Possible scoring ranges from 0 to 100, the greater the score the greater the functional capability, lower the score the increase chances of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Director — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No